CLINICAL TRIAL: NCT07214545
Title: Phase IIa Clinical Trial of External Trigeminal Nerve Stimulation for Autistic Children With Attention Deficit/Hyperactivity Disorder
Brief Title: External Trigeminal Nerve Stimulation for Children With ASD + ADHD to Reduce Elevated Symptoms
Acronym: eTNS CARES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, James T McCracken, M.D., Deputy Vice Chair for Research-Child, Moghadam Family Distinguished Professor, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 25-44041
Record Dates: First submitted 2025-09-11; First posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Attention Deficit Disorder With Hyperactivity (ADHD); Autism Spectrum Disorder (ASD)
Keywords: eTNS; external trigeminal nerve stimulation; eTNS CARES
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active eTNS Device (Active Comparator)
  Interventions: Device: Trigeminal Nerve Stimulation
- Sham eTNS Device (Sham Comparator)
  Interventions: Device: Sham Trigeminal Nerve Stimulation

INTERVENTIONS:
Device: Trigeminal Nerve Stimulation — This intervention is expected to have an effect following a treatment period of 6 weeks.
  Arms: Active eTNS Device
Device: Sham Trigeminal Nerve Stimulation — This intervention is NOT expected to have an effect following a treatment period of 6 weeks.
  Arms: Sham eTNS Device

SUMMARY:
The goal of this clinical trial is to learn if external trigeminal nerve stimulation (eTNS) works to treat ADHD symptoms in children on the autism spectrum (ASD). It will also learn about the efficacy and tolerability of the eTNS device. The main questions it aims to answer are:

* Does eTNS reduce ADHD symptoms?
* Does eTNS improve core and associated features of ASD?

Participation spans 8-12 weeks and includes:

* 4-5 in-person visits
* 4 brief virtual check-ins
* Nightly use of the eTNS device with a small sticky patch applied to child's forehead
* Randomized assignment (those who start with the sham device may try the active device later)

ELIGIBILITY:
Inclusion Criteria:

* Confirmed clinician diagnosis of ASD according to DSM-5 criteria, corroborated by prior testing (or obtained in study screening) with the Autism Diagnostic Observation Schedule (ADOS) with or without the Autism Diagnostic Interview-Revised (ADI-R)
* IQ > 70 as corroborated by prior testing (or obtained in study screening) with the Wechsler Abbreviated Scale of Intelligence Scale (WASI)
* Confirmed diagnosis of ADHD according to DSM-5 criteria with minimum ADHD-RS score of > 24
* Stable on current medications for a minimum of 4 weeks before baseline
* Ability to complete protocol testing
* Both the child participant and their primary caregiver must be fluent in English (speaking, reading, and understanding), as the questionnaires and assessment tools used in this study have been validated only in English.

Exclusion Criteria:

* Current major depression, history of psychosis, bipolar disorder, elevated risk of self-harm
* History of moderate to severe coarse brain injury
* Active medical illness expected to interfere with study assessments
* Presence of implanted stimulator (e.g., vagal nerve stimulator)
* Active dermatologic condition likely to interfere with eTNS electrode wearability
* Sleep disorder likely to interfere with nightly eTNS in the opinion of the study physician
* Inability to communicate discomfort or pain
* Current and anticipated continued use of antipsychotic or stimulant medication

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-10-06 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in ADHD Symptoms | Baseline to end of treatment at 6 weeks
  Examine the efficacy of external Trigeminal Nerve Stimulation (eTNS) in reducing ADHD symptoms as measured by the Attention-Deficit/Hyperactivity Disorder Rating Scale-5 (ADHD-RS-5; range 0-54), where higher scores indicate worse symptoms.

SECONDARY OUTCOMES:
Change in Social Responsiveness | Baseline to end of treatment at 6 weeks
  Examine changes in social communication and related behaviors as measured by the Social Responsiveness Scale, Second Edition, Short Form (SRS-2-SF; range 0-48), where higher scores indicate worse impairment.
Change in Restricted and Repetitive Behaviors | Baseline to end of treatment at 6 weeks
  Examine changes in restricted and repetitive behaviors as measured by the Repetitive Behavior Scale-Revised (RBS-R; range 0-129), where higher scores indicate more severe repetitive behaviors.
Change in Sleep Quality | Baseline to end of treatment at 6 weeks
  Examine changes in sleep quality as measured by the Children's Sleep Habits Questionnaire (CSHQ; range 33-99), where higher scores indicate poorer sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- UCSF Nancy Friend Pritzker Psychiatry Building, San Francisco, California, United States